CLINICAL TRIAL: NCT01277783
Title: ALternate Site Cardiac ReSYNChronization Study
Brief Title: ALternate Site Cardiac ReSYNChronization (ALSYNC) Study
Acronym: ALSYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSYNC
Record Dates: First submitted 2011-01-11; First posted 2011-01-17 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endocardial Left Ventricular pacing (Experimental): All patients will undergo the intervention, and are followed at 1, 3, 6, and 12 months (minimum) and biannually thereafter until 1 year after enrollment of the last patient.
  Interventions: Device: Endocardial Left Ventricular pacing

INTERVENTIONS:
Device: Endocardial Left Ventricular pacing — Subjects receive an endocardial LV lead placement via superior approach using Medtronic Model 3830 lead and Medtronic Model 6227ATS deflectable delivery catheter and Medtronic Model 6248HS, 6248JL, or 6248JS delivery catheter, using trans esophageal echo (TEE) or intra-cardiac echo (ICE) to guide the procedure.

SUMMARY:
The ALternate site cardiac reSYNChronization (ALSYNC) study, a non-comparative, prospective, non-randomized, multi-national clinical investigation.

The purpose of this clinical investigation is to evaluate the safety and performance of the investigational atrial transseptal endocardial LV lead delivery system and the implant procedure for delivering the SelectSecure® Model 3830 lead into the Left Ventricle via a superior approach, and to evaluate the performance of the SelectSecure® Model 3830 lead in the Left Ventricle.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) reduces mortality and the risk of heart failure decompensation and improves quality of life in indicated patients. However, many do not benefit due to failure to deliver the left ventricular (LV) lead via coronary sinus (5-10%) or lack of symptomatic improvement (30-40%).

The purpose of the ALSYNC Study was to evaluate the feasibility and safety of LV endocardial (LVE) pacing using a Model 3830 lead implanted by a novel pectoral atrial transseptal lead delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Resynchronization Therapy candidate/recipient with:
* Failed Cardiac Resynchronization Therapy implant or required CRT replacement without viable access to Coronary sinus or,
* Sub-optimal Coronary sinus anatomy per investigator discretion or,
* Worsened or unchanged clinical status after Cardiac Resynchronization Therapy implant
* Patients able and willing to take optimal Vitamin K antagonist therapy (International Normalized Ratio (INR) of 2-4)
* Patients willing to sign and date the Patient Informed Consent form
* Patients 18 years of age or older
* Patients able and willing to comply with the protocol, and is expected to remain available for follow-up visits

Exclusion Criteria:

* Patients having contraindications to Vitamin K antagonist therapy
* Patients contraindicated for < 100 micrograms beclomethasone dipropionate
* Patients unable to tolerate an urgent thoracotomy
* Documented (previous) ischemic or hemorrhagic stroke
* Patients with known previous atrial septal defect closure, or history of mural thrombus that has not been resolved
* Patients with documented atrial fibrillation AND increased stroke risk as determined by the Congestive Heart Failure, Hypertension, Age(2), Diabetes, Stroke(2), Vascular disease, Age, and Sex Category (CHA2DS2-VASc) Score of equal to or greater than 5
* Patients with unstable angina pectoris or who have had an acute myocardial infarct within the past 30 days
* Patients with known atrial septum defect (ASD) and/or left superior vena cava
* Patient with known internal carotid artery stenosis of greater than 50%
* Patients diagnosed with peripheral artery disease that are expected to undergo stenting within the next three months
* Patients who have had a Coronary artery bypass graft or stent within the past three months
* Patients with history of mitral or aortic valve repair or replacement
* Post heart transplant patients (patients waiting for heart transplant are allowed in the study)
* Patients currently undergoing dialysis treatment
* Patients with ongoing chemotherapy and radiation therapy that may have an effect on cardiac function
* Patients with ongoing Adverse Events from a previous Left Ventricle lead implant attempt
* Patients enrolled in any concurrent drug and/or device study that may confound the results of this study
* Patients who are not expected to survive more than twelve months
* Patients with exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor John Morgan, MD, Principal Investigator — Spire Southampton Hospital
Locations (18):
- Belgium (2):
  - AZ Sint-Jan - Campus Sint-Jan, Bruges
  - Centre Hospitalier Regional de la Citadelle, Liège
- Canada (2):
  - Saint Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre - University Campus, London, Ontario
- France (5):
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Bordeaux
  - CHU Grenoble Hôpital Michalon, Grenoble
  - Infirmerie Protestante de Lyon, Lyon
  - Nouvelles Cliniques Nantaises, Nantes
  - Hôpital Pontchaillou - CHU de Rennes, Rennes
- Semmelweis Egyetem AOK, Budapest, Hungary
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant' Orsola - Malpighi, Bologna
  - Presidio Ospedaliero Alessandro Manzoni, Lecco
  - Azienda Complesso Ospedaliero San Filippo Neri Ospedale San Filippo Neri, Roma
- Academisch Ziekenhuis Maastricht (AZM), Maastricht, Netherlands
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Golden Jubilee National Hospital, Glasgow
  - University College London Hospitals NHS Foundation Trust - The Heart Hospital, London
  - Southampton General Hospital, Southhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biffi M, Defaye P, Jais P, Ruffa F, Leclercq C, Gras D, Yang Z, Gerritse B, Ziacchi M, Morgan JM; ALSYNC Investigators. Benefits of left ventricular endocardial pacing comparing failed implants and prior non-responders to conventional cardiac resynchronization therapy: A subanalysis from the ALSYNC study. Int J Cardiol. 2018 May 15;259:88-93. doi: 10.1016/j.ijcard.2018.01.030. PMID 29579617
- [Derived] Morgan JM, Biffi M, Geller L, Leclercq C, Ruffa F, Tung S, Defaye P, Yang Z, Gerritse B, van Ginneken M, Yee R, Jais P; ALSYNC Investigators. ALternate Site Cardiac ResYNChronization (ALSYNC): a prospective and multicentre study of left ventricular endocardial pacing for cardiac resynchronization therapy. Eur Heart J. 2016 Jul 14;37(27):2118-27. doi: 10.1093/eurheartj/ehv723. Epub 2016 Jan 18. PMID 26787437

RESULTS

PARTICIPANT FLOW:
Groups:
- LV Endocardial Lead: subjects receive an endocardial LV lead placement via superior approach using Medtronic Model 3830 lead and Medtronic Model 6227ATS deflectable delivery catheter and Medtronic Model 6248HS, 6248JL, or 6248JS delivery catheter and guidance of TEE or ICE.
  Medtronic Model 6227ATS deflectable delivery catheter: Endocardial Left Ventricular pacing lead delivery
  Medtronic Model 6248HS, 6248JL, or 6248JS delivery catheter: Endocardial Left Ventricular pacing lead delivery
  Medtronic Model 3830: Endocardial Left Ventricular pacing
Period: Overall Study
Arm/Group | LV Endocardial Lead
Started | 138
Completed | 138
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects meeting eligibility criteria are included in the baseline analysis population. 2 subjects were not included from the overall number of subjects that completed the study because they had a major eligibility violation (both had left superior vena cava).
Groups:
- Left Ventricular Endocardial Pacing: All enrolled patients were scheduled to receive a CRT implantation with endocardial LV lead
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 136
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 66 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender (male) | 106
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — Classification of symptoms:
  Class I=No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea.
  Class II=Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  Class III=Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV=Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA Class I | 4
    NYHA Class II | 29
    NYHA Class III | 93
    NYHA Class IV | 10
Atrial Fibrillation [Count of Participants; unit: Participants] — Number of subjects that have Atrial Fibrillation at baseline
  Participants | 68
Left Bundle Branch Block (LBBB) [Count of Participants; unit: Participants] — Number of subjects that have LBBB at baseline
  Participants | 94
QRS duration [Mean (Standard Deviation); unit: milliseconds (ms)] — The duration in milliseconds (ms) of the QRS complex in the subject's electrocardiogram at baseline.
  milliseconds (ms) | 165 (32)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percentage] — The percentage of blood leaving the heart each time it contracts
  percentage | 29 (9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free From Lead, Delivery System and Implant Related Complications.
Description: Adverse events were reviewed by an independent Adverse Event Adjudication Committee. Events classified as complication related to the LV endocardial lead, the investigational delivery system or the implant procedure contribute to the outcome. The percentage of patients free from such complication at 6 months after the procedure was estimated using the Kaplan-Meier method and is reported with the corresponding 95% confidence interval.
Time Frame: 6 months
Population: The Analysis cohort (132) includes the Baseline cohort (136) (Enrolled patients (138), excluding patients exited for eligibility violation without implant attempt and patients removed for major eligibility violation (2)), excluding patients that did not have implant attempt (4).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | LV Endocardial Lead
Number analyzed (Participants) | 132
percentage of patients | 82.2 [75.6 to 88.8]

2. Secondary Outcome: Implant Success
Description: Number of participants with a successful implant of Model 3830 lead.
Time Frame: Implant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LV Endocardial Lead
Number analyzed (Participants) | 132
Participants | 118

3. Secondary Outcome: Number of Questionnaires Reporting None of the Handling and Implant Characteristics as Poor
Description: Questionaires were collected for each LV lead implant attempt, reattempt, and LV lead modification. To evaluate the ease of positioning of the Model 3830 lead and the Models 6227ATS and 6248HS, JS, JL catheters, a rating scale of Poor, Fair, Good, Very good, and Excellent was used for each of the ten questions on the questionnaire. Outcome reports the number of questionnaires where no single question was answered with Poor.
Time Frame: Implant
Population: Participants analyzed are those in the Analysis cohort as described before (132). The unit of analysis is a questionnaire for each attempted Model 3820 lead implant (139). In 7 cases their was a repeat procedure (reported as repeat implant attempt or system modification).
Measure: Count of Units; unit: questionnaire
Units Other Than Participants: questionnaire
Arm/Group | LV Endocardial Lead
Number analyzed (Participants) | 132
Number analyzed (questionnaire) | 139
questionnaire | 75

4. Secondary Outcome: Bipolar Sensing Amplitude of the Model 3830 Lead in the LV at 12 Months
Description: Sensing amplitude measurement was taken with the implanted device at the 12 month follow-up visit.
Time Frame: 12 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 24 patients had a missing 12-months follow-up visit and 5 had a missing R-wave amplitude measurement
Measure: Mean (Standard Deviation); unit: Bipolar Sensing Amplitude in milliVolts
Groups:
- Left Ventricular Endocardial Pacing: subjects receive an endocardial LV lead placement via superior approach using Medtronic Model 3830 lead and Medtronic Model 6227ATS deflectable delivery catheter and Medtronic Model 6248HS, 6248JL, or 6248JS delivery catheter and guidance of TEE or ICE.
  Medtronic Model 6227ATS deflectable delivery catheter: Endocardial Left Ventricular pacing lead delivery Medtronic Model 6248HS, 6248JL, or 6248JS delivery catheter: Endocardial Left Ventricular pacing lead delivery Medtronic Model 3830: Endocardial Left Ventricular pacing
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 89
Bipolar Sensing Amplitude in milliVolts | 11 (6.4)

5. Secondary Outcome: Bipolar Pacing Threshold of the Model 3830 Lead in the LV at 12 Months
Description: Bipolar measurement of Model 3830 lead voltage threshold at 0.4ms pulse width using the implanted device at the 12 month visit
Time Frame: 12 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 24 patients had a missing 12-months follow-up visit and 4 had a missing bipolar pacing threshold measurement
Measure: Mean (Standard Deviation); unit: Bipolar LV pacing threshold in Volts
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 90
Bipolar LV pacing threshold in Volts | 0.84 (0.27)

6. Secondary Outcome: Bipolar Pacing Impedance of the Model 3830 Lead in the LV at 12 Months
Description: Measurement of Impedance of the Model 3830 Lead in the LV using the implanted device at the 12 month visit
Time Frame: 12 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 24 patients had a missing 12-months follow-up visit and 3 had a missing impedance measurement
Measure: Mean (Standard Deviation); unit: Bipolar LV Pacing Impedance in Ohms
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 91
Bipolar LV Pacing Impedance in Ohms | 596 (80)

7. Secondary Outcome: Subjects With 1 Class of NYHA Improvement From Baseline to 6 Months
Description: NYHA Class change was evaluated between baseline and the 6 months visit. Reported are the subjects with at least 1 class improvement from baseline to 6 months
Time Frame: baseline and 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 13 patients had a missing 6-months follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 105
Participants | 62

8. Secondary Outcome: Distance Walked at 6 Minute Hall Walk at the 12 Month Visit
Description: Distance walked at the 6 minute hall walk test at the 12 month visit
Time Frame: 12 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 24 patients had a missing 12-months follow-up visit, and 18 did not complete the test.
Measure: Mean (Standard Deviation); unit: Distance walked in meters
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 76
Distance walked in meters | 391 (147)

9. Secondary Outcome: Percent Change in Left Ventricular Ejection Fraction From Baseline to 6 Months
Description: Percent change in Left Ventricular Ejection Fraction (LVEF) was measured from baseline to 6 months
Time Frame: baseline and 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 18 patients had a missing LVEF measurement at baseline and/or 6 months.
Measure: Mean (Standard Deviation); unit: Percent change in LVEF
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 100
Percent change in LVEF | 36.1 (12.0)

10. Secondary Outcome: Milliliters Change in Left Ventricular End-Systolic Volume at 6 Months
Description: Milliliters change in Left Ventricular End-Systolic Volume (LVESV) from baseline to 6 months
Time Frame: 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 27 patients had a missing LVESV measurement at baseline and/or 6 months.
Measure: Mean (Standard Deviation); unit: LVESV change in milliliters
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 91
LVESV change in milliliters | 121 (74)

11. Secondary Outcome: Millimeters Change in Left Ventricular End-Diastolic Diameter From Baseline to 6 Months
Description: Millimeters change in Left Ventricular End-Diastolic Diameter (LVEDD) from baseline to 6 months
Time Frame: baseline and 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 17 patients had a missing LVEDD measurement at baseline and/or 6 months.
Measure: Mean (Standard Deviation); unit: millimeters change in LVEDD
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 101
millimeters change in LVEDD | 63.7 (9.9)

12. Secondary Outcome: Number of Subjects With Mitral Regurgitation Improvement of at Least One Class From Baseline to 6 Months
Description: Reported is the number of patients with at least one class improvement from baseline to 6 months
Time Frame: baseline and 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 16 patients had a missing MR measurement at baseline and/or 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 102
Participants | 33

13. Secondary Outcome: Change in (NT-pro)BNP Levels From Baseline to 6 Months
Description: Change in either Brain Natriuretic Peptide (BNP) or N-Terminal-prohormone BNP (NT-proBNP) levels from baseline to 6 months
Time Frame: baseline and 6 months
Population: Of the 118 patients that were successfully implanted with the Model 3830 lead in the LV, 22 patients had a missing (NTpro)BNP measurement at baseline and/or 6 months.
Measure: Mean (Standard Deviation); unit: change in picograms per milliliter
Arm/Group | Left Ventricular Endocardial Pacing
Number analyzed (Participants) | 86
change in picograms per milliliter
  BNP: number analyzed (Participants) | 31
  BNP | 444 (587)
  NT-proBNP: number analyzed (Participants) | 55
  NT-proBNP | 2554 (3485)

ADVERSE EVENTS:
Time Frame: Serious adverse events are reported with onset between the start of the LV endocardial implant procedure and the end of follow-up, which was after 17.3 months on average.
Description: Serious adverse events are reported for the 132 patients that had an attempt to implant an endocardial LV lead. Implantation was successful for 118 patients.
Arm/Group | Left Ventricular Endocardial Pacing
All-Cause Mortality (participants affected / at risk) | 23/132
Serious Adverse Events (participants affected / at risk) | 86/132
Other Adverse Events (participants affected / at risk) | 49/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Ventricular Endocardial Pacing (N=132)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 3
Atrial thrombosis (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 30
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Electromechanical dissociation (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 4
Macular oedema (Eye disorders) | 1
Retinal artery thrombosis (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Cardiac failure (General disorders) | 1
Chest pain (General disorders) | 1
Implant site haematoma (General disorders) | 8
Presyncope (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1
Device dislocation (Injury, poisoning and procedural complications) | 1
Device lead damage (Injury, poisoning and procedural complications) | 2
Device migration (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Implant site reaction (Injury, poisoning and procedural complications) | 1
Lead dislodgement (Injury, poisoning and procedural complications) | 6
Wound dehiscence (Injury, poisoning and procedural complications) | 1
International normalised ratio decreased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Cognitive disorder (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 7
Device psychogenic complication (Psychiatric disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Cardiac failure (Surgical and medical procedures) | 1
Extrusion of device (Surgical and medical procedures) | 1
Peripheral revascularisation (Surgical and medical procedures) | 1
Arterial disorder (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Implant site haematoma (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Ventricular Endocardial Pacing (N=132)
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 2
Atrial tachycardia (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 7
Intracardiac thrombus (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Metamorphopsia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal disorder (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Implant site fibrosis (General disorders) | 1
Implant site haematoma (General disorders) | 8
Oedema (General disorders) | 1
Bronchitis (Infections and infestations) | 5
Catheter related infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 1
Inappropriate device therapy (Injury, poisoning and procedural complications) | 3
Lead dislodgement (Injury, poisoning and procedural complications) | 2
International normalised ratio increased (Investigations) | 1
Troponin (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Vascular dementia (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Implant site haematoma (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No